CLINICAL TRIAL: NCT04994210
Title: Safety and Efficacy of Sintilimab(S) in Combination With Histone Deacetylase Inhibitor (Chidamide, C) in Newly Diagnosed Extranodal Natural Killer Cell/T-cell Lymphoma(EN): A Single-arm, Multicenter Phase II Study(SCENT-2)
Brief Title: Sintilimab in Combination With Chidamide in Newly Diagnosed ENKTCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huiqiang Huang, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCENT-2
Record Dates: First submitted 2021-07-22; First posted 2021-08-06 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Safety and Efficacy
Keywords: Sintilimab; Chidamide; refractory and relapsed; Extranodal natural killer cell/T-cell lymphoma
MeSH Terms: conditions — Recurrence | interventions — sintilimab; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab+Chidamide (Experimental): Sintilimab：200mg(fixed dosage), ivd, qd, q21d Chidamide: 30mg,biw,continued oral
  Interventions: Drug: Sintilimab; Drug: Chidamide

INTERVENTIONS:
Drug: Sintilimab — 1. To evaluate the short-term objective efficacy of sintilimab combined with chidamide in the treatment of newly diagnosed ENKTCL patients
  2. To evaluate the long-term efficacy and safety of sintilimab combined with chidmide in the treatment of newly diagnosed ENKTCL patients.
  3. Exploring biomarkers that may have predictive effects.
  Other Names: Tyvyt®
Drug: Chidamide — 1. To evaluate the short-term objective efficacy of sintilimab combined with chidamide in the treatment of newly diagnosed ENKTCL patients
  2. To evaluate the long-term efficacy and safety of sintilimab combined with chidmide in the treatment of newly diagnosed ENKTCL patients.
  3. Exploring biomarkers that may have predictive effects.
  Other Names: Epidaza

SUMMARY:
ENKTL is a highly aggressive NHL with a higher incidence in Asia. L-asparaginase containing chemotherapy regimens are the standard first-line treatment with apparently toxicities. In 2020 ASH, the investigators reported Sintilimab(anti-PD-1 antibody) plus Chidamide(an oral subtype-selective HDACi) yielded effective antitumor activity, durable response in patients with relapsed or refractory ENKTL(SCENT trial. Abstracts 644). The investigators next conducted a exploratory study to investigated the safety and efficacy of Sintilimab plus Chidamide(SC) for patients with newly diagnosed ENKTL(SCENT-2 trial).

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in clinical research; fully understand and know the research and sign the Informed Consent Form (ICF); willing to follow and have the ability to complete all trial procedures;
2. Aged 18-80 years old male or female;
3. Extranodal NK/T-cell lymphoma confirmed by histopathology examination;
4. Untreated,without any anti-lymphoma treatment;
5. Paraffin tissue specimens or fresh puncture tissue specimens are available;
6. Eastern cooperative oncology group score: 0-2;
7. Estimated survival ≥ 12 months;
8. There must be at least one evaluate able or measurable lesion that meets the lymphoma response to immunomodulatory therapy criteria (LYRIC) [evaluable lesion: 18F-fluorodeoxyglucose/Positron Emission Tomography (18FDG/PET) examination showing increased lymph node or extranodal uptake (higher than liver) and PET and/or computed tomography (Computed Tomography) CT) features are consistent with lymphoma findings; lesions can be measured: nodular lesions > 15mm or extranodal lesions > 10mm (if the only measurable lesion has received radiotherapy in the past, there must be evidence of radiological progress after radiotherapy), and accompanied by increased 18FDG uptake). Except for this, there is no measurable increase in diffuse 18FDG uptake in the liver;
9. Adequate organ and bone marrow function, no severe hematopoietic dysfunction, cardiac, pulmonary, liver, kidney, thyroid dysfunction and immune deficiency (no blood transfusion, granulocyte colony stimulating factor or other medical support was received within 14 days prior to the use of the research drug): 1) The absolute value of neutrophils (>1.0×10^9/L); 2) platelet count (> 75×10^9/L); 3) Hemoglobin (> 9 g/dL); 4) Upper Limit Normal (ULN) or creatinine clearance rate (>40 mL/min) of serum creatinine (<1.5 times normal value upper limit) (estimated by Cockcroft-Gault formula); 5) Serum total bilirubin < 1.5 times ULN; 6) Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) = 2.5 times ULN; 7) Coagulation function: International Normalized Ratio (INR) = 1.5 times ULN; Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT) = 1.5 times ULN (unless the subject is receiving anticoagulant therapy and PT and APTT are using anticoagulant therapy at screening time). Within the expected range; 8) Thyrotropin (TSH) or free thyroxine (FT4) or free triiodothyronine (FT3) were all within the normal range (+10%);
10. There was no evidence that subjects had difficulty breathing at rest, and the measured value of pulse oximetry at rest was more than 92%;
11. Participants must pass a pulmonary function test (PFT) to confirm that forced expiratory volume (FEV1)/forced vital capacity (FVC) in the first second is more than 60%, unless it is a large mediastinal mass caused by lymphoma that cannot meet this standard; carbon monoxide diffusion (DLCO), FEV1 and FVC are all above 50% of the predicted value; all PFT results must be obtained within four weeks before the first administration;
12. Women of Childbearing Potential (WOBCP) must undergo a serum pregnancy test within seven days before the first medication and the results are negative. WOBCP or men and their WOBCP partners should agree to take effective contraceptive measures from the signing of ICF until six months after the last dose of the research drug is used

Exclusion Criteria:

1. Invasive natural killer cell leukemia;
2. Hemophagocytic syndrome;
3. Primary central nervous system lymphoma or secondary central nervous system involvement;
4. Relapsed or refractory ENKTL, accpeted any anti-ENKTL treatment;
5. Received organ transplantation in the past;
6. Participating in other clinical studies or planning to start this study is less than 4 weeks from the end of the previous clinical study;
7. Patients with active autoimmune diseases requiring systematic treatment in the past two years (hormone replacement therapy is not considered systematic treatment, such as type I diabetes mellitus, hypothyroidism requiring only thyroxine replacement therapy, adrenocortical dysfunction or pituitary dysfunction requiring only physiological doses of glucocorticoid replacement therapy); Patients with autoimmune diseases who do not require systematic treatment within two years can be enrolled;
8. Begin the study on subjects requiring systemic glucocorticoid therapy or other immunosuppressive therapy for a given condition within 14 days before treatment [allowing subjects to use local, ocular, intra-articular, intranasal and inhaled glucocorticoid therapy (with very low systemic absorption); and allowing short-term (< 7 days) glucocorticoid prophylaxis (e.g., contrast agent overdose) Sensitivity) or for the treatment of non-autoimmune diseases (e.g. delayed hypersensitivity caused by contact allergens);
9. In the past five years, patients with other malignant tumors have undergone radical treatment, except for basal cell carcinoma of skin, squamous cell carcinoma of skin, carcinoma in situ of breast and carcinoma in situ of cervix;
10. Start the study and receive Chinese herbal medicine or Chinese patent medicine treatment within 7 days before treatment;
11. Begin research on live vaccination (except influenza attenuated vaccine) within 28 days before treatment;
12. History of human immunodeficiency virus (HIV) infection and/or patients with acquired immunodeficiency syndrome are known;
13. Patients with active hepatitis B or active hepatitis C. Patients who are positive for hepatitis B Surface Antigen (HBsAg) or hepatitis C Virus (HCV) antibodies at screening stage must pass further detection of hepatitis B Virus (HBV) DNA titer (no more than 2500 copies/mL or 500 IU/mL) and HCV RNA (no more than the lower limit of the detection method) in the row. In addition to active hepatitis B or hepatitis C infections requiring treatment, group trials can be conducted. Hepatitis B carriers, stable hepatitis B (DNA titer should not be higher than 2500 copies/mL or 500 IU/mL) after drug treatment, and cured hepatitis C patients can be enrolled in the group;
14. Patients with active pulmonary tuberculosis;
15. Start studying any active infections requiring systemic anti-infective treatment within 14 days of treatment;
16. Pregnant or lactating women;
17. People with known history of alcoholism or drug abuse;
18. Have uncontrollable complications, including but not limited to symptomatic congestive heart failure, uncontrollable hypertension, unstable angina, active peptic ulcer or hemorrhagic diseases;
19. History of interstitial lung disease or non-infectious pneumonia. Subjects who had previously had non-infectious pneumonia caused by drugs or radiation but had no symptoms were allowed to enter the group;
20. The QTcF interval is more than 450 msec, unless it is secondary to bundle branch block;
21. Past psychiatric history; incapacitated or restricted;
22. According to the researchers'judgment, patients' underlying condition may increase their risk of receiving research drug treatment, or confuse their judgment on toxic reactions;
23. Other researchers consider it unsuitable for patients to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) after end of treatment | up to 24 months
  Assessed by the lymphoma response to immunomodulatory therapy criteria (LYRIC)
Complete response rate (CRR) after end of treatment | up to 24 months
  Assessed by the lymphoma response to immunomodulatory therapy criteria (LYRIC)
Partial response rate (PRR) after end of treatment | up to 24 months
  Assessed by the lymphoma response to immunomodulatory therapy criteria (LYRIC)

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Time Frame: up to 36 months
  PFS is defined as the time from the treatment date to the date of disease progression per the RECIL 2017 Response Criteria for Malignant Lymphoma or death regardless of cause.
Overall Survival (OS) | up to 36 months
  OS is defined as the time from treatment to the date of death.
Duration of Response (DOR) | up to 36 months
  Among participants who experience an objective response, DOR is defined as the date of their first objective response (which is subsequently confirmed) to disease progression per the the lymphoma response to immunomodulatory therapy criteria (LYRIC) or death regardless of cause.
Time to disease response (TTR) | up to 36 months
  Among participants who experience an objective response, TTR is defined as the date of their first administration to the day of their first objective response (which is subsequently confirmed) per the RECIL 2017 Response Criteria for Malignant Lymphoma.
Time to progression (TTP) | Up to 36 months
  Among all participants, TTP is defined as the date of their first administration to the day of disease progression per the RECIL 2017 Response Criteria for Malignant Lymphoma or death regardless of cause.
The frequency of adverse events (adverse events, AEs) and serious adverse events (SAEs) | Up to 36 months
  An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAE were defined as AEs with onset during the treatment period or that are a consequence of a pre-existing condition that has worsened since baseline.
Objective response rate (ORR) after sintilimab plus chidamide | up to 24 months
  Assessed by the lymphoma response to immunomodulatory therapy criteria (LYRIC)
Complete response rate (CRR) after sintilimab plus chidamide | up to 24 months
  Assessed by the lymphoma response to immunomodulatory therapy criteria (LYRIC)
Partial response rate (PRR) after sintilimab plus chidamide | up to 24 months
  Assessed by the lymphoma response to immunomodulatory therapy criteria (LYRIC)

CONTACTS AND LOCATIONS:
Locations (1):
- SunYat-sen university cancer center, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided